CLINICAL TRIAL: NCT01904318
Title: A Dose Block-randomized, Doubled, Placebo-controlled, Single Dose, Dose-escalation Clinical Phase I Study to Evaluate the Safety, Pharmacokinetics and Food
Brief Title: A Phase I Study of IDP-73152 Mesylate in Health Male Volunteer
Acronym: PDF inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID-PDF-70-1
Record Dates: First submitted 2013-07-16; First posted 2013-07-22 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: male; Phase I; A dose block-randomized; Double-blinded; Placebo controlled; Single Dose; dose Escalation; IDP-73152 mesylate; Food Effect; Pharmacokinetics; health male volunteer; PDF inhibitor
MeSH Terms: interventions — IDP-73152

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- IDP-73152 mesylate 40 mg (Experimental)
  Interventions: Drug: IDP-73152 mesylate 40 mg
- IDP-73152 mesylate 80 mg (Experimental)
  Interventions: Drug: IDP-73152 mesylate 80 mg
- IDP-73152 mesylate 160 mg (Experimental)
  Interventions: Drug: IDP-73152 mesylate 160 mg
- IDP-73152 mesylate 320 mg (Experimental)
  Interventions: Drug: IDP-73152 mesylate 320 mg
- IDP-73152 mesylate 640 mg (Experimental)
  Interventions: Drug: IDP-73152 mesylate 640 mg
- IDP-73152 mesylate 1280 mg (Experimental)
  Interventions: Drug: IDP-73152 mesylate 1280 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IDP-73152 mesylate 40 mg — IDP-73152 mesylate 40 mg single dose administration
  Arms: IDP-73152 mesylate 40 mg
Drug: IDP-73152 mesylate 80 mg — IDP-73152 mesylate 80 mg single dose administration
  Arms: IDP-73152 mesylate 80 mg
Drug: IDP-73152 mesylate 160 mg — IDP-73152 mesylate 160 mg single dose administration
  Arms: IDP-73152 mesylate 160 mg
Drug: IDP-73152 mesylate 320 mg — IDP-73152 mesylate 320 mg single dose administration
  Arms: IDP-73152 mesylate 320 mg
Drug: IDP-73152 mesylate 640 mg — IDP-73152 mesylate 640 mg single dose administration
  Arms: IDP-73152 mesylate 640 mg
Drug: IDP-73152 mesylate 1280 mg — IDP-73152 mesylate 1280 mg single dose administration
  Arms: IDP-73152 mesylate 1280 mg
Drug: Placebo — Placebo single dose administration
  Arms: Placebo

SUMMARY:
A dose block-randomized, double-blinded, placebo-controlled, single dose, dose-escalation clinical phase I study to evaluate the safety, pharmacokinetics and food effect of IDP-73152 mesylate after oral administration in healthy male volunteer

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-50 years inclusive, at screening visit.
* 55kg ≤ Body weight ≤90kg and body mass index (BMI) between 18.0 - 25.0 kg/m2.
* Subject does not have congenital or chronic disease and is without pathologic symptom or finding on medical exam.
* Subject was determined eligible according to the results of clinical laboratory tests like serum test, hematologic test, blood chemistry test, urine test etc. and vital signs, electrocardiography, physical exam etc. performed during the screening exam.
* Subject decided to participate voluntarily and gave written Informed consent to comply with the instructions after listening to and fully understanding the detailed explanation about this trial.

Exclusion Criteria:

* Subject has clinically significant liver, kidney, neurologic, immunologic, respiratory, endocrine disease or hematologic•oncologic disease, cardiovascular disease or psychiatric disease (mood disorder, compulsive disorder etc.) or such medical history (including subject with hepatitis virus in case of liver disease).
* Subject has history of gastrointestinal disease (such as Crohn's disease, ulcer, acute or chronic pancreatitis etc.) or gastrointestinal surgery (except simple appendectomy or hernia operation) that can affect the absorption of the study drug.
* Subject has hypersensitivity reaction to drug (aspirin, antibiotics etc.) or history of clinically significant hypersensitivity reaction.
* Specific laboratory values at screening including: AST(SGOT) and/or ALT > 1.25 times the upper limit of normal; QTc > 430 ms or clinical significance of abnormal electrocardiographic patterns.
* Uncontrolled hypertension defined as sustained systolic blood pressure (SBP) < 90 mmHg or > 150 mmHg or diastolic BP (DBP) < 60 mmHg or > 110 mmHg at screening evaluation.
* History of recent tobacco abuse in the past 3 months.
* Subject took any prescribed drug or oriental medicine within 2 weeks prior to the first medication or any over-the-counter (OTC) drug or vitamins within 1 week prior to the first medication (however, the subject can be included if other criteria are met according to the discretion of the investigator).
* Use of an investigational drug or treatment in past 2months
* Subject donated whole blood within 2 months prior to the first medication or apheresis within 1 month prior to the first medication or received blood transfusion within 1 month prior to the first medication.
* Subject continually drinks (in excess of 21 units/week, 1 unit = 10 g of pure alcohol) or cannot abstain from drinking through the study period.
* History of recent tobacco abuse (within 3 months)
* Subject took grapefruit/caffeine-containing food within 3 days prior to the first medication, or cannot abstain from taking during the hospitalization period.
* Subject was judged not to be eligible according to the discretion of the investigator for other reasons.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Vital signs | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 days
Electrocardiography | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 days
Clinical laboratory tests | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 days
Physical exam | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 day
Adverse event | participants will be followed for the duration of hospital stay and post study visit, an expected average of 10 days

SECONDARY OUTCOMES:
Cmax, Cmax/D, AUClast, AUClast/D, AUCinf, AUCinf/D of IDP-73152 mesylate | Pre-dose (0 h), Post-dose (0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10,12, 24, 36, 48 h)
Tmax, T1/2, CL/F, CLr of IDP-73152 mesylate | Pre-dose (0 h), Post-dose (0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10,12, 24, 36, 48 h)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Sang you, MD, PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Jongno-gu, Seoul, South Korea